CLINICAL TRIAL: NCT04762745
Title: Department of Hematologic Oncology, Sun Yat-sen University Cancer Center, Guangzhou, China
Brief Title: The Efficacy and Safety of Pomalidomide and Bendamustine With Dexamethasone in Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hua Wang, Associate professor of Department of Hematological Oncology, Sun Yat-sen University Cancer Center, Guangzhou, China, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRMM-01
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Relapsed, Refractory, Multiple Myeloma
Keywords: pomalidomide, bendamustine, multiple myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — pomalidomide; Bendamustine Hydrochloride; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase I, Cohort 1 (Experimental): The combination of bendamustine, 60mg/m2, with pomalidomide and dexamethasone will be administrated in 6 relapsed or refractory multiple myeloma patients for 1 cycle. If dose limiting toxicity (DLT) is observed in 2 or more of the six patients at the same dosing level while DLT is observed in only 1 or none of the 6 patients at the dosing level immediately below it, then the lower dosing level will be defined as the maximum tolerated dose (MTD).
  Interventions: Drug: Pomalidomide; Drug: Bendamustine; Drug: Dexamethasone
- Phase I, Cohort 2 (Experimental): The combination of bendamustine, 70mg/m2, with pomalidomide and dexamethasone will be administrated in 6 relapsed or refractory multiple myeloma patients for 1 cycle. If dose limiting toxicity (DLT) is observed in 2 or more of the six patients at the same dosing level while DLT is observed in only 1 or none of the 6 patients at the dosing level immediately below it, then the lower dosing level will be defined as the maximum tolerated dose (MTD).
  Interventions: Drug: Pomalidomide; Drug: Bendamustine; Drug: Dexamethasone
- Phase I, Cohort 3 (Experimental): The combination of bendamustine, 80mg/m2, with pomalidomide and dexamethasone will be administrated in 6 relapsed or refractory multiple myeloma patients for 1 cycle. If dose limiting toxicity (DLT) is observed in 2 or more of the six patients at the same dosing level while DLT is observed in only 1 or none of the 6 patients at the dosing level immediately below it, then the lower dosing level will be defined as the maximum tolerated dose (MTD).
  Interventions: Drug: Pomalidomide; Drug: Bendamustine; Drug: Dexamethasone
- Phase II (Experimental): The combination of MTD dosage of bendamustine with pomalidomide and dexamethasone will be administrated in an expanded relapsed or refractory multiple myeloma cohorts for 8 cycles, then under the combination of pomalidomide and dexamethasone as maintenance therapy until progression or intolerable toxicities.
  Interventions: Drug: Pomalidomide; Drug: Bendamustine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide( Anyue®, Chia Tai TIANQING, China), 4mg, orally(PO), d1-21, 28d/cycle, 1cycle.
  Other Names: Pomalidomide( Anyue®, Chia Tai TIANQING, China)
  Arms: Phase I, Cohort 1
Drug: Bendamustine — Bendamustine( Leweixin®, Chia Tai TIANQING, China), 60mg/m2/d, intravenously(IV), d1-2, 28d/cycle, 1 cycle.
  Other Names: Bendamustine( Leweixin®, Chia Tai TIANQING, China)
  Arms: Phase I, Cohort 1
Drug: Dexamethasone — Dexamethasone, 40mg, PO or IV, d1, 8, 15, 22, 28d/cycle, 1 cycle.
  Arms: Phase I, Cohort 1
Drug: Pomalidomide — Pomalidomide( Anyue®, Chia Tai TIANQING, China), 4mg, orally(PO), d1-21, 28d/cycle, 1cycle.
  Other Names: Pomalidomide( Anyue®, Chia Tai TIANQING, China)
  Arms: Phase I, Cohort 2
Drug: Bendamustine — Bendamustine( Leweixin®, Chia Tai TIANQING, China), 70mg/m2/d, intravenously(IV), d1-2, 28d/cycle, 1 cycle.
  Other Names: Bendamustine( Leweixin®, Chia Tai TIANQING, China)
  Arms: Phase I, Cohort 2
Drug: Dexamethasone — Dexamethasone, 40mg, PO or IV, d1, 8, 15, 22, 28d/cycle, 1 cycle.
  Arms: Phase I, Cohort 2
Drug: Pomalidomide — Pomalidomide( Anyue®, Chia Tai TIANQING, China), 4mg, orally(PO), d1-21, 28d/cycle, 1cycle.
  Other Names: Pomalidomide( Anyue®, Chia Tai TIANQING, China)
  Arms: Phase I, Cohort 3
Drug: Bendamustine — Bendamustine( Leweixin®, Chia Tai TIANQING, China), 70mg/m2/d, intravenously(IV), d1-2, 28d/cycle, 1 cycle.
  Other Names: Bendamustine( Leweixin®, Chia Tai TIANQING, China)
  Arms: Phase I, Cohort 3
Drug: Dexamethasone — Dexamethasone, 40mg, PO or IV, d1, 8, 15, 22, 28d/cycle, 1 cycle.
  Arms: Phase I, Cohort 3
Drug: Pomalidomide — Pomalidomide( Anyue®, Chia Tai TIANQING, China), 4mg, orally(PO), d1-21, 28d/cycle, 8 cycles. Then pomalidomide( Anyue®, Chia Tai TIANQING, China), 4mg, orally(PO), d1-21, 28d/cycle until progression or intolerable toxicities.
  Other Names: Pomalidomide( Anyue®, Chia Tai TIANQING, China)
  Arms: Phase II
Drug: Bendamustine — Bendamustine( Leweixin®, Chia Tai TIANQING, China), 70mg/m2/d, intravenously(IV), d1-2, 28d/cycle, 8 cycles.
  Other Names: Bendamustine( Leweixin®, Chia Tai TIANQING, China)
  Arms: Phase II
Drug: Dexamethasone — Dexamethasone, 40mg, PO or IV, d1, 8, 15, 22, 28d/cycle, 8 cycles. Then dexamethasone, 40mg, PO or IV, d1, 8, 15, 22, 28d/cycle until progression or intolerable toxicities.
  Arms: Phase II

SUMMARY:
To explore the efficacy and safety of pomalidomide and bendamustine with dexamethasone in relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
The trial has two parts: firstly, to explore the maximum tolerated dosage(MTD) of bendamustine in the combination of pomalidomide and dexamethasone in relapsed or refractory multiple myeloma; secondly, to find out efficacy and safety of pomalidomide and bendamustine with dexamethasone in relapsed or refractory multiple myeloma in an expanded cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75, no gender limitations.
* Ability of contraception during the experiment, no matter if they have suffered from infertility.
* Relapsed or refractory to prior lenalidomide or/and bortezomib(either in combination or sequential)therapy (i.e. history of progression on therapy or within 60 days after completion)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2, life expectancy of more than 6 months.
* Measurable disease:

Serum M protein > 10 g/L or Urine M protein ≥200 mg/24 hr or Elevated Free Light Chain per International Myeloma Working Group (IMWG) criteria, and abnormal ratio.

* Absolute neutrophil count (ANC) >1.0 x 109/L or >1.0 x 109/L due to granulocyte/macrophage colony stimulating factor (GCSF and GMCSF), or if >50% marrow involvement, there is no limitations
* Platelet count >50.0 x 109/L or if >50% marrow involvement, there is no limitations.
* Total bilirubin ≤ 2.0mg/dL, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the upper limit of normal.
* Serum creatinine ≤2.0 mg/dL or creatinine clearance ≥60ml/min.
* Agree to take anticoagulant drugs, included but not limited to aspirin.
* Agree to sign the informed consent form.

Exclusion Criteria:

* Patients with known sensitivity to pomalidomide or bendamustine or dexamethasone and their accessories.
* Patients with primary systemic amyloidosis or monoclonal gammopathy of undetermined significance or smoldering multiple myeloma.
* Patients with active new thrombosis or disagree to take anticoagulant drugs, included but not limited to aspirin.
* Active treatment or intervention for other malignancy or need active treatment within 4 weeks of starting study treatment. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Central nervous system involvement.
* Systemic treatment with immunodepressants or steroids.
* Ongoing or active systemic infection, active hepatitis B virus infect, active hepatitis C infection, or known human immunodeficiency virus (HIV) positive
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure(NT-Pro-BNP≥1800pg/mL), unstable angina, or myocardial infarction within the past 6 months.
* Infection requiring systemic antibiotic therapy or other serious infection.
* Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens. Psychiatric illness/social situation that would limit compliance with study requirements.
* Under other clinical trial procedures.
* Female patients who are lactating or pregnant.
* Other patients not appropriate for the trial in the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At the end of Cycle 8 in Phase II (each cycle is 28 days)
  The number of patients achieving partial response (PR), very good partial response (VGPR), complete response (CR) or stringent complete response (sCR) after 8 cycles in phase II.
  sCR = CR as defined in Primary Outcome measure 2 plus normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
  CR- Negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
  VGPR = Serum and urine M-protein detectable by immunofixation but not on electrophoresis or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 h.
  PR- > 50% reduction of serum M-protein and urine M-protein by >90% or to < 200 mg/24 h In addition, if present at baseline, a > 50% reduction in the size of soft tissue plasmacytomas is also required.

SECONDARY OUTCOMES:
Complete response(CR) and stringent complete response(sCR) rate | At the end of Cycle 8 in Phase II (each cycle is 28 days)
  The CR and sCR rate after 8 cycles in phase II.
  CR- Negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
  sCR = CR as defined in Primary Outcome measure 2 plus normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Progression free survival(PFS) | Through study completion, up to 2 years
  The time relapsed for patients between initiation of study therapy and either disease progression or death
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, up to 2 years
  Number of participants with treatment-related adverse events during the study period as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Please Select, China

IPD SHARING:
Plan to Share IPD: No